CLINICAL TRIAL: NCT00762528
Title: Compare Anti-inflammatory Dentifrices
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-1107-INF-ECU-FP
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2012-04-03 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-08

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Triclosan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total Toothpaste (Active Comparator): Triclosan/Copolymer/fluoride toothpaste
  Interventions: Drug: Triclosan/Copolymer/fluoride toothpaste
- Fluoride toothpaste (Placebo Comparator): sodium monofluorophosphate toothpaste
  Interventions: Drug: Sodium monofluorophosphate toothpaste

INTERVENTIONS:
Drug: Triclosan/Copolymer/fluoride toothpaste — Twice daily usage
  Other Names: Toothpaste includes triclosan/fluoride/co-polymer (Total)
  Arms: Total Toothpaste
Drug: Sodium monofluorophosphate toothpaste — Twice daily usage
  Other Names: fluoride only toothpaste
  Arms: Fluoride toothpaste

SUMMARY:
Plaque induced gingivitis

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be adult males or females 18 to 60 years old
* Subjects must be able and willing to follow study procedures and instructions
* Subjects must have read, understood and signed an informed consent form
* Subjects must have generalized, moderate plaque-associated gingivitis as determined by the Investigator or designee during the screening examination
* Subjects must present with at least 20 teeth in the functional dentition, excluding third molars
* Each subject must have at least four teeth with probing depths of 4-5 mm and at least 30% of sites bleeding to gentle probing

Exclusion Criteria:

* Subjects who have chronically used (i.e., two weeks or more) Total (Triclosan/Copolymer) dentifrice within 6 months prior to enrollment
* Subjects with gross oral pathology, including widespread caries or chronic neglect, extensive restoration, pre-existing gross plaque and calculus, or soft or hard tissue tumor of the oral cavity
* Subjects with periodontitis as indicated by periodontal pocketing 6 mm at screening
* Subjects with a history of early onset periodontitis or acute necrotizing ulcerative gingivitis
* Subjects with concomitant endodontic or periodontal therapy other than prophylaxis within 6 months prior to enrollment
* Subjects with orthodontic appliances or removable partial dentures
* Subjects chronically treated (two weeks or more) with any medication known to affect inflammation or periodontal status or (aspirin, nonsteroidal anti-inflammatory drugs, steroids, statins, phenytoin, calcium antagonists, cyclosporin and coumadin) within one month of the screening examination. All other medications for chronic medical conditions should be initiated at least three months prior to enrollment
* Subjects who currently smoke or who report using tobacco products within one year of screening.
* Subjects who have been treated with antibiotics for medical or dental reasons within 3 months prior to enrollment
* Subjects having clinically significant or unstable organic disease; subjects having compromised healing potential such as those with diabetes mellitus or connective tissue disorders; subjects having heart murmurs, histories of rheumatic fever, valvular disease or prosthetic joint replacement necessitating antibiotic prophylaxis
* Female subjects who report being pregnant or lactating, or female subjects who are of childbearing potential and who report not using hormonal or barrier methods of birth control (oral or parenteral contraceptives, diaphragm plus spermicide, condoms)
* Subjects who use hormonal contraceptives must have started the method 30 days prior to the screening examination.
* Subjects with active infectious diseases such as hepatitis, human immunodeficiency virus or Tuberculosis
* Subjects diagnosed with human immunodeficiency virus (HIV) or subjects that are immunocompromised as determined by the Investigator
* Medical condition which precludes not eating/drinking for approximately 8 hours.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara G Grossi, DDS, Principal Investigator
Locations (1):
- East Carolina University, Brody School of Medicine, Greenville, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subject recruitment will be completed by the PI at the clinical site.
Pre-assignment Details: Subjects are screened for plaque, bleeding and gingivitis scores before being assigned to any Study Treatment. Study Treatment randomization is balanced across the two treatment groups and is accomplished by stratification of subjects by gender (male & female) and baseline gingivitis (GI) scores.
Period: Overall Study
Arm/Group | Total Toothpaste | Fluoride Toothpaste
Started | 24 | 25
Completed | 24 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Toothpaste | Fluoride Toothpaste | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 25 | 49
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (10.7) | 29.2 (9.6) | 28.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 12 | 13 | 25
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: Gingival Index (GI)
Description: Gingival Index(GI)recorded on scale of 0-3 detailed below:
  0=normal gingiva, 1=Mild inflammation(slight change in color, slight edema)no bleeding on palpation,2=Moderate inflammation(redness,edema,glazing)bleeding upon probing, 3=Severe inflammation(marked redness,edema)ulceration & tendency to spontaneously bleed
Time Frame: 29 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Toothpaste | Fluoride Toothpaste
Number analyzed (Participants) | 24 | 25
units on a scale | 1.04 (0.22) | 1.01 (0.19)
Statistical Analysis 1: Comparison: Total Toothpaste vs Fluoride Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.05, ANOVA

2. Primary Outcome: Prostaglandin E2 (PGE2)
Description: Inflammatory biomarker found in gingival crevicular fluid (GCF). Higher Levels found in GCF may be a factor in tissue destruction as seen in periodontal disease. All GCF samples are collected onto filter paper strips (Pro Flow, Inc.) and the volume determined by Periotron 8000. Samples were placed in cryovial and labelled, then place into liquid nitrogen and stored at -180°C until analysis.
Time Frame: 29 days
Measure: Log Mean (Standard Deviation); unit: pg/µl
Arm/Group | Total Toothpaste | Fluoride Toothpaste
Number analyzed (Participants) | 24 | 25
pg/µl | 5.8 (2.7) | 5.2 (3)
Statistical Analysis 1: Comparison: Total Toothpaste vs Fluoride Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.05, ANOVA

3. Primary Outcome: Interleukin - 1 Beta (IL-ß)
Description: Inflammatory biomarkers found in gingival crevicular fluid (GCF) that may be a factor in oral tissue destruction as seen in periodontal disease. All GCF samples are collected onto filter paper strips (Pro Flow, Inc.) and the volume determined by Periotron 8000. Samples were placed in cryovial and labelled, then place into liquid nitrogen and stored at -180°C until analysis.
Time Frame: 29 days
Measure: Log Mean (Standard Deviation); unit: pg/µl
Arm/Group | Total Toothpaste | Fluoride Toothpaste
Number analyzed (Participants) | 24 | 25
pg/µl | 6.9 (0.8) | 6.6 (1.2)
Statistical Analysis 1: Comparison: Total Toothpaste vs Fluoride Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.05, ANOVA

4. Secondary Outcome: Dental Plaque Index (PI)
Description: measurement of supragingival dental plaque on scale of 0-3. 0=No plaque in gingival area,1=a film of plaque adhering to the free gingival margin and the adjacent tooth,2=Moderate accumulation of soft deposits within the gingival pocket and on the gingival margin and/or adjacent tooth-visible by the naked eye, 3=Abundance of soft matter within the gingival pocket and/or gingival margin and adjacent tooth surfaces.
Time Frame: 29 days
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Total Toothpaste | Fluoride Toothpaste
Number analyzed (Participants) | 24 | 25
Units on a scale | 1.69 (0.30) | 1.65 (0.35)
Statistical Analysis 1: Comparison: Total Toothpaste vs Fluoride Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.05, ANOVA

5. Secondary Outcome: Bleeding on Probing (BOP)
Description: Presence or absence of bleeding to manual probing as a dichotomous variable as follows: 0 = No bleeding within 10 seconds after probing, 1 = Bleeding within 10 seconds after probing.
Time Frame: 29 days
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Total Toothpaste | Fluoride Toothpaste
Number analyzed (Participants) | 24 | 25
Units on a scale | 0.24 (0.10) | 0.26 (0.12)
Statistical Analysis 1: Comparison: Total Toothpaste vs Fluoride Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.05, ANOVA

6. Primary Outcome: Interleukin-6 (IL-6)
Description: as for outcome 2
Time Frame: 29 days
Measure: Log Mean (Standard Deviation); unit: pg/µl
Arm/Group | Total Toothpaste | Fluoride Toothpaste
Number analyzed (Participants) | 24 | 25
pg/µl | 2.8 (0.7) | 2.7 (0.6)
Statistical Analysis 1: Comparison: Total Toothpaste vs Fluoride Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.05, ANOVA

7. Primary Outcome: Nuclear Factor Kappa B Ligand (RANK-L)
Description: Receptor activator found in gingival crevicular fluid (GCF). Presence in GCF may indicate tissue damage as seen in periodontal disease. All GCF samples are collected onto filter paper strips (Pro Flow, Inc.) and the volume determined by Periotron 8000. Samples were placed in cryovial and labelled, then place into liquid nitrogen and stored at -180°C until analysis.
Time Frame: 29 days
Measure: Log Mean (Standard Deviation); unit: pg/µl
Arm/Group | Total Toothpaste | Fluoride Toothpaste
Number analyzed (Participants) | 24 | 25
pg/µl | 4.5 (0.9) | 4.4 (1)
Statistical Analysis 1: Comparison: Total Toothpaste vs Fluoride Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.05, ANOVA

8. Primary Outcome: 8-iso-prostaglandinF2α (8-iso-PGF2α)
Description: Inflammatory biomarker found in gingival crevicular fluid (GCF). Presence in GCF may indicate tissue damage as seen in periodontal disease. All GCF samples are collected onto filter paper strips (Pro Flow, Inc.) and the volume determined by Periotron 8000. Samples were placed in cryovial and labelled, then place into liquid nitrogen and stored at -180°C until analysis.
Time Frame: 29 days
Measure: Log Mean (Standard Deviation); unit: pg/µl
Arm/Group | Total Toothpaste | Fluoride Toothpaste
Number analyzed (Participants) | 24 | 25
pg/µl | 14.2 (3.8) | 15.2 (1.6)
Statistical Analysis 1: Comparison: Total Toothpaste vs Fluoride Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 29 days
Arm/Group | Total Toothpaste | Fluoride Toothpaste
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 1/24 | 6/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Toothpaste (N=24) | Fluoride Toothpaste (N=25)
Teeth Sensitive to cold (General disorders) | 0 (0) | 2 (2) — 2 subjects reported tooth sensitivity to cold.
Oral Irritation (General disorders) | 0 (0) | 1 (1) — subject reported oral irritation
chest cold, upper respiratory infection (General disorders) | 1 (1) | 1 (1) — 2 subjects reported having a cold
Pulled muscle in back (General disorders) | 0 (0) | 1 (1) — subject reported having a pulled muscle in their back.
Fever, chills & sore throat (General disorders) | 0 (0) | 1 (1) — subject reported experiencing a fever, chills and sore throat.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less